CLINICAL TRIAL: NCT05432245
Title: A Prospective, Open, Multicenter Clinical Trial Evaluating the Efficacy and Safety of MINIject Combined With Cataract Surgery in Patients With POAG Uncontrolled by Topical Hypotensive Medications and Operable Age-related Cataract Diagnosis
Brief Title: MINIject Implantation Combined With Cataract Surgery in Patients With POAG and Cataract
Acronym: STAR-VI
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: iSTAR Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STAR VI
Record Dates: First submitted 2022-06-16; First posted 2022-06-27 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Primary Open-angle Glaucoma; Cataract
Keywords: Primary Open-angle Glaucoma (POAG); Cataract; Intra Ocular Pressure (IOP) reduction; Glaucoma Drainage Device; Minimally Invasive Glaucoma Surgery (MIGS); Supraciliary space; Combined procedure (POAG and phacoemulsification)
MeSH Terms: conditions — Glaucoma, Open-Angle; Cataract

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment group (Experimental)
  Interventions: Device: Phacoemulsification combined with minimally invasive glaucoma surgery (MIGS)

INTERVENTIONS:
Device: Phacoemulsification combined with minimally invasive glaucoma surgery (MIGS) — The cataract surgery will be performed first and if successful, only then will the MINIject be placed into supraciliary space.

SUMMARY:
The study will assess safety and performance of MINIject implant in patients with open-angle glaucoma uncontrolled by topical hypotensive medications in conjunction with cataract surgery.

DETAILED DESCRIPTION:
The study aims to evaluate the safety and efficacy of the MINIject in the reduction of intraocular pressure (IOP) in patients with primary open-angle glaucoma (POAG) in conjunction with cataract surgery. The cataract surgery will be performed first and if successful, only then will the MINIject be placed.

Patients will be followed for 2 years after the date of their implantation. Standard ophthalmologic assessments including measurement of intraocular pressure, fundus examination, ocular imaging, assessment of any untoward ocular events etc. will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of primary open angle glaucoma (POAG) in the study eye
* Operable age-related cataract eligible for phacoemulsification surgery with Intraocular Lens (IOL) implantation
* Glaucoma not adequately controlled with at least one topical hypotensive medication(s), unless the patient has an allergy / intolerance to a medication
* Patient must provide written informed consent to participate

Exclusion Criteria:

* Known or suspected allergy or hypersensitivity to medical silicone
* Allergy to fluorescein
* Presence of silicone oil in the study eye
* Individuals under tutorship or trusteeship
* Patient has a condition such that his / her ability to provide personal informed consent is compromised

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-01-18 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Proportion of study eyes achieving ≥ 20% reduction in diurnal IOP | 6 months
  Proportion of study eyes achieving ≥ 20% reduction in diurnal IOP from baseline to 6 months follow-up, with or without IOP lowering medications

CONTACTS AND LOCATIONS:
Overall Officials: Zubair Hussain, PhD, Study Director — iSTAR Medical
Locations (4):
- Panama Eye Center, Panama City, Panama
- Hospital Clínico San Carlos, Madrid, Spain
- United Kingdom (2):
  - East Suffolk and North Essex NHS Foundation Trust - Colchester General Hospital, Colchester, Essex
  - Princess Alexandra Eye Pavilion, Edinburgh

IPD SHARING:
Plan to Share IPD: No